CLINICAL TRIAL: NCT00661765
Title: A Phase I, Open-Label, Randomized, Single Dose, Cross Over Study to Estimate the Relative Bioavailability of a Varenicline (CP-526,555) Transdermal Delivery System to the Chantix Immediate Release Tablet Formulation in Adult Smokers
Brief Title: A Single Dose Study Investigating the Absorption and Elimination as Well as the Tolerability of Varenicline Transdermal Delivery System (e.g., a Patch) as Compared to Oral Varenicline in Adult Smokers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A3051071
Record Dates: First submitted 2008-04-14; First posted 2008-04-18 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Smoking Cessation
Keywords: varenicline bioavailability transdermal smoking cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chantix immediate release tablet formulation (Active Comparator)
  Interventions: Drug: varenicline tartrate
- Varenicline transdermal delivery system (Experimental)
  Interventions: Drug: varenicline free base

INTERVENTIONS:
Drug: varenicline tartrate — Single dose of 2.0 mg oral Chantix (varenicline) immediate release tablet formulation
  Other Names: varenicline, Chantix, Champix
  Arms: Chantix immediate release tablet formulation
Drug: varenicline free base — A single 2.0 mg dose of varenicline transdermal delivery system applied to the skin for a 24 hour period.
  Other Names: varenicline
  Arms: Varenicline transdermal delivery system

SUMMARY:
1. To evaluate the absorption and elimination of varenicline Formulation A transdermal delivery system [TDS (patch)] compared to varenicline immediate release tablet (CHANTIX®).
2. To evaluate the adhesion of the varenicline Formulation A patch.
3. To evaluate the safety and tolerability of a single application of the varenicline patch and a single oral dose of the varenicline immediate release tablet (CHANTIX®).

ELIGIBILITY:
Inclusion Criteria:

* healthy adult smokers

Exclusion Criteria:

* Significant blood, kidney, lung, gastrointestinal, heart, liver, psychiatric, or neurologic disease
* Illegal drug usage

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Rating Scale for Adhesive Residue (e.g., assesses how well the transdermal delivery system remains adhered to subject's skin) | 24 hours per Arm
Rating Scale for Assessment of Application Site Dermal-Erythema, Edema, and Irritation (assesses skin irritation associated with varenicline transdermal delivery system) | 6 days per Arm
Pharmacokinetic endpoints: plasma varenicline area under the curve (AUClast and AUCinf), maximum plasma concentration (Cmax), terminal half-life (t 1/2) and time of maximum plasma concentration (Tmax) | 6 days per Arm

SECONDARY OUTCOMES:
Assessment of Adhesidue/Cold Flow Assessment (assesses extent of adhesive residue which remains on the skin at application site as well as the adhesive flow beyond the application site border | 24 hours per Arm
Evaluation of adverse events (including the visual analog scale for nausea), safety laboratory testing, electrocardiogram, vital signs | 6 days per Arm

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Fargo, North Dakota, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051071&StudyName=A%20single%20dose%20study%20investigating%20the%20absorption%20and%20elimination%20as%20well%20as%20the%20tolerability%20of%20%20varenicline%20transdermal%20delivery%20system